CLINICAL TRIAL: NCT07182968
Title: Cultural Adaptation, Validity, and Reliability of the Turkish Version of the Patient Assessment of Skin Thickness in the Upper Limb - PASTUL Questionnaire
Brief Title: Cultural Adaptation, Validity, and Reliability of the Turkish Version of The PASTUL Questionnaire
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Other Study IDs: SBA 24/531
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis (SSc); Systemic Sclerosis (Scleroderma); Scleroderma (Limited and Diffuse); Patient Perspective
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Systemic sclerosis
  Interventions: Other: Questionnaire study

INTERVENTIONS:
Other: Questionnaire study — Questionnaire application

SUMMARY:
The Patient Self-Assessment of Skin Thickness in Upper Limb (PASTUL) questionnaire was developed to enable patients to assess skin thickness in systemic sclerosis (SSc) physically and has been validated for reliability and validity, as it correlates with the modified Rodnan Skin Score (mRSS), which rheumatologists assess. Thus, it has been demonstrated to be an applicable and easy approach for assessing skin thickness in SSc patients through patient-reported measurements. This study aimed to develop a Turkish version of the PASTUL questionnaire and to provide for its use in the Turkish population.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with scleroderma,
* Individuals aged 18 years and older

Exclusion Criteria:

* Advanced heart/lung/liver/kidney disease, neurological disease, and malignancies
* Individuals who are unwilling to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08-04 (Estimated)

PRIMARY OUTCOMES:
Patient Self-Assessment of Skin Thickness in Upper Limb (PASTUL) Questionnaire | Two weeks
  The PASTUL survey is a simple assessment by the patient of the skin in eight areas of the upper extremities as normal, mildly, moderately, or severely thickened, corresponding to the mRSS assessment. The assessment score is consistent with the mRSS (0-3). A high score indicates increased skin thickness

SECONDARY OUTCOMES:
Scleroderma Health Assessment Questionnaire (SHAQ) | Two weeks
  It was developed by adding five questions to the HAQ regarding Raynaud's phenomenon, digital ulcers, gastrointestinal, pulmonary, and general scleroderma symptoms, to be rated on a 15 cm line. The SHAQ total score ranges from 0 to 3. A high score indicates low functionality.
Cognitive Exercise Therapy Approach-Biopsychosocial Questionnaire (BETY-BQ) | Two weeks
  It was standardized as a biopsychosocial assessment tool and is scored using a 5-point Likert scale, with each item rated from 0 to 4 points. A high total score on the 30-item scale indicates a high level of biopsychosocial impact.
Short Form-36 (SF-36) | Two weeks
  It will be used to determine an individual's quality of life levels. Each sub-parameter is scored between 0 and 100 points, with a high score indicating good health status. The SF-36 scale has eight sub-parameters: general health perception, physical function, social function, pain, mental health, role difficulty due to physical reasons, role difficulty due to emotional reasons, and vitality. It contains 11 questions consisting of a total of 36 items.
Modified Rodnan skin score (MRSS) | Two weeks
  A pediatric and adult rheumatologist assessed it. The MRSS evaluates skin thickening in 17 body regions, graded from 0 (normal) to 3 (severe skin thickening). The total score ranges from 0 to 51, with increased scores indicating poor skin involvement.
Modified Hand Mobility in Scleroderma Test (mHAMIS) | Two weeks
  It is a functional test developed specifically for scleroderma to assess an individual's hand function. It evaluates four specific hand movements (finger flexion, finger extension, finger abduction, and dorsal extension). Scores range from 0 (normal) to 3 (complete failure) for each movement, with a total score ranging from 0 to 12.
Scleroderma Skin Patient-Reported Outcomes (SSPRO) Questionnaire | Two weeks
  It assesses the impact of skin involvement on quality of life. The 18-item measure consists of 4 categories: physical effect (PE), emotional effect (EE), social effect (SE), and physical limitation (PL). Each item is scored on a scale ranging from no impairment (0 points) to severe impairment (6 points), with a total score of 108. A lower score indicates a much better quality of life.
Cochin Hand Function Scale | Two weeks
  It consists of 18 questions related to daily activities. Each question is scored on a questionnaire of 0 (no difficulty) to 5 (impossible), and the total score ranges from 0 to 90. A total CHFS score of 26 or higher is considered to indicate hand function limitation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No